CLINICAL TRIAL: NCT05006209
Title: Comparison of One-visit Root Canal Treatment Using Chlorhexidine as a Final Irrigant and Conventional Two-visit Root Canal Treatment
Brief Title: One-visit Root Canal Treatment Using Chlorhexidine as a Final Irrigant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Seniha Miçooğulları Kurt, Principle investigator, Asst. Assoc. Dr, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: one-visit root canal treatment
Record Dates: First submitted 2021-07-24; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Root Canal Infection
Keywords: chlorhexidine; one visit root canal treatment
MeSH Terms: interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One visit root canal treatment with CHX (Active Comparator): The teeth were treated in one-visit (OV) root canal treatment. Final root canal irrigation was performed with 5% EDTA, followed by 2.5% NaOCl and received an additional final rinse with 2% CHX before obturation.
  Interventions: Other: One visit root canal treatment
- Two visit root canal treatment with CH (Active Comparator): The teeth were treated in two visit (TV) root canal treatment. After completion of root canal instrumentation, calcium hydroxide (CH) paste was placed into the root canal. In second visit, all root canals were irrigated with 5% EDTA followed by 2.5% NaOCl before obturation.
  Interventions: Other: Two visit root canal treatment

INTERVENTIONS:
Other: One visit root canal treatment
  Other Names: CHX
  Arms: One visit root canal treatment with CHX
Other: Two visit root canal treatment
  Other Names: Calcium hydroxide
  Arms: Two visit root canal treatment with CH

SUMMARY:
A hundred asymptomatic molar teeth with periapical lesions were treated in single versus multiple visit root canal treatment. Half of the teeth were randomly assigned to the one-visit (OV) group and received an additional final rinse with 2% CHX before obturation. The other teeth were treated in two visits (TV) with calcium hydroxide dressing. All patients were recalled and investigated clinically and radiographically for 48 months

DETAILED DESCRIPTION:
The aim of the study was to evaluate the radiographic evidence of periapical healing in teeth with apical periodontitis treated in a single visit with an additional final irrigation using 2% chlorhexidine and to compare the results with conventional multiple-visit root canal treatment (RCT) with an intracanal calcium hydroxide dressing as a control group. 100 asymptomatic molar teeth with periapical lesions were treated using engine-driven nickel-titanium (NiTi) instrumentation with 2.5% sodium hypochlorite (NaOCl) and 5% ethylenediaminetetraacetic acid (EDTA) as irrigants. Half of the teeth were randomly assigned to the one-visit (OV) group and received an additional final rinse with 2% chlorhexidine (CHX) before obturation. The other teeth were treated in two visits (TV), after completion of root canal instrumentation calcium hydroxide paste was placed into the root canal and root canal obturation was performed in second visit. All patients were recalled and investigated clinically and radiographically for 48 months. Changes in apical bone density indicating radiographic healing were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* with a non-contributory medical history,
* mature molar teeth with periapical lesions,
* diagnosed as asymptomatic apical periodontitis

Exclusion Criteria:

* clinical symptoms, drainage,
* more than 5 mm loss of periodontal attachment,
* previous endodontic treatment,
* non-restorable tooth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical healing according to presence of clinical symptoms | 12 months
  All patients were called for follow up visits. The clinical healing was determined by examining clinical symptoms including presence of pain, tenderness to percussion and palpation, presence of sinus tract or swelling, and mobility. If one of these symptoms occurs, it is considered as failure..
Clinical healing according to presence of clinical symptoms | 24 months
  All patients were called for follow up visits. The clinical healing was determined by examining clinical symptoms including presence of pain, tenderness to percussion and palpation, presence of sinus tract or swelling, and mobility.If one of these symptoms occurs, it is considered as failure..
Clinical healing according to presence of clinical symptoms | 48 months
  All patients were called for follow up visits. The clinical healing was determined by examining clinical symptoms including presence of pain, tenderness to percussion and palpation, presence of sinus tract or swelling, and mobility.If one of these symptoms occurs, it is considered as failure..
Changes in the size and the PAI score of the periapical lesion | 12 months
  The rate of radiographic healing of the periapical lesion. Follow-up visits were performed for all patients in order to evaluate radiographic status. Changes in apical bone density indicating radiographic healing was assessed using Periapical Index (PAI)(Orstavik 1986) as the scoring system.
Changes in the size and the PAI score of the periapical lesion | 24 months
  The rate of radiographic healing of the periapical lesion. Follow-up visits were performed for all patients in order to evaluate radiographic status. Changes in apical bone density indicating radiographic healing was assessed using Periapical Index (PAI)(Orstavik 1986) as the scoring system.
Changes in the size and the PAI score of the periapical lesion | 48 months
  The rate of radiographic healing of the periapical lesion. Follow-up visits were performed for all patients in order to evaluate radiographic status. Changes in apical bone density indicating radiographic healing was assessed using Periapical Index (PAI)(Orstavik 1986) as the scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Seniha Miçooğulları Kurt, Principal Investigator — Ege University Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Micoogullari Kurt S, Caliskan MK. Efficacy of chlorhexidine as a final irrigant in one-visit root canal treatment: a prospective comparative study. Int Endod J. 2018 Oct;51(10):1069-1076. doi: 10.1111/iej.12931. Epub 2018 Apr 23. PMID 29603299
- [Background] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729
- [Background] Siqueira JF Jr, Rocas IN. Optimising single-visit disinfection with supplementary approaches: a quest for predictability. Aust Endod J. 2011 Dec;37(3):92-8. doi: 10.1111/j.1747-4477.2011.00334.x. PMID 22117714